CLINICAL TRIAL: NCT06930898
Title: Improving Breast Health Knowledge Among Women Using a Gamified Metaverse-Based Platform: A Randomized Controlled Trial
Brief Title: Improving Breast Health Knowledge Among Women Using a Gamified Metaverse-Based Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Mammo2025-RCT01; UMREC_3967 (Other: University of Malaya Research Ethics Committee)
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Health Education; Breast Neoplasms
Keywords: Gamification; Health Education; Breast Cancer Awareness; Metaverse; Women's Health; Digital Health Literacy
MeSH Terms: conditions — Health Education; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to one of two parallel groups: a gamified version of the Mammoverse metaverse-based platform or a non-gamified version containing the same educational content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gamified Metaverse Education (Experimental): Participants in this group used the Mammoverse platform with gamified features, including story-based missions, interactive tasks, point-based rewards, achievement badges, and virtual incentives. The educational content was delivered through immersive scenarios to enhance engagement and motivation in learning about breast health.
  Interventions: Behavioral: Gamified Mammoverse Platform
- Non-Gamified Metaverse Education (Active Comparator): Participants in this group accessed the Mammoverse platform without any gamified features. The virtual environment delivered identical breast health educational content, but without tasks, points, rewards, badges, or narrative elements.
  Interventions: Behavioral: Standard Mammoverse Platform

INTERVENTIONS:
Behavioral: Gamified Mammoverse Platform — A gamified, metaverse-based platform delivering breast health education through story-based tasks, interactive challenges, points, rewards, badges, and virtual incentives.
  Arms: Gamified Metaverse Education
Behavioral: Standard Mammoverse Platform — A non-gamified version of the Mammoverse platform that provides the same breast health educational content.
  Arms: Non-Gamified Metaverse Education

SUMMARY:
This randomized controlled trial aimed to evaluate the effectiveness of Mammoverse, a gamified metaverse-based educational platform, in improving breast health knowledge among women in China. Participants were randomly assigned to either a gamified or non-gamified version of the platform. Both groups received identical educational content, but only the gamified group experienced interactive game elements such as avatars, progress feedback, and rewards. Knowledge was assessed at baseline, immediately post-intervention, and at 4-week follow-up. The study found that the gamified platform significantly improved knowledge retention and participant engagement compared to the non-gamified version.

This ClinicalTrials.gov registration reflects only the randomized controlled trial (RCT) portion of a broader mixed-methods study that was approved by the University of Malaya Research Ethics Committee (Ref: UM.TNC2/UMREC_3967). The full study protocol includes three methodological approaches, and this registration pertains specifically to the RCT component involving the Mammoverse platform. Other study components are not included in this registration.

DETAILED DESCRIPTION:
Mammoverse is a 3D metaverse environment designed to promote breast health knowledge through immersive and interactive learning. The gamified version included user avatars, badges, tasks, and personalized feedback to increase motivation and engagement. The study recruited 72 women aged 18 and above, and used a pre-post-follow-up design. Outcome measures were based on an adapted 18-item Breast Health Literacy Questionnaire. The trial was conducted entirely online, with ethics approval from the University of Malaya Research Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18 years and above
* Able to read and understand Chinese
* Access to a digital device and stable internet connection
* Willing to provide informed consent

Exclusion Criteria:

* Cognitive impairment or mental health condition that affects participation
* Inability to complete the full intervention and follow-up sessions
* Incomplete baseline assessment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Change in Breast Health Knowledge Score from Baseline to 4 Weeks Post-Intervention | Baseline and 4 weeks post-intervention
  Assessed using an 18-item adapted Breast Health Literacy Questionnaire. Scores range from 0 to 18, with higher scores indicating greater knowledge. Main comparison is between baseline and 4-week follow-up.

SECONDARY OUTCOMES:
Change in Breast Health Knowledge Score from Baseline to Immediately Post-Intervention | Baseline and immediately post-intervention
  Same questionnaire used to assess immediate knowledge gain after the intervention.

OTHER OUTCOMES:
Knowledge Retention from Immediately Post-Intervention to 4 Weeks Post | Immediately post-intervention and 4 weeks post-intervention
  Change in knowledge scores to evaluate retention over 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Li, PhD(c), Principal Investigator — University of Malaya
Locations (2):
- Online Recruitment - Hangzhou, Zhejiang, China, Hangzhou, Zhejiang, China
- University of Malaya, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li R, Kahn SM, Duan B, Wong SY. Gamified Versus Non-gamified Metaverse Learning for Breast Health Knowledge in Women: Randomized Controlled Trial. JMIR Serious Games. 2026 Jan 6. doi: 10.2196/75318. Online ahead of print. PMID 41499212